CLINICAL TRIAL: NCT06793085
Title: Assessment of the Concentrations of Pro- and Anti-inflammatory Cytokines and Their Association With the Metabolic Profile of Women With PCOS
Brief Title: Pro- and Anti-inflammatory Cytokines in PCOS
Status: Recruiting | Type: Observational
Sponsor: Jagiellonian University (Other)
Responsible Party: Principal Investigator, Iwona Magdalena Gawron, PhD, MD, Principal Investigator, Jagiellonian University
Other Study IDs: 1072.6120.44.2024-2
Record Dates: First submitted 2025-01-20; First posted 2025-01-27 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Reproductive Age; PCOS (Polycystic Ovary Syndrome)
Keywords: menstrual disorders; chronic inflammation; insulin resistance; metabolic syndrome; Polycystic Ovary Syndrome
MeSH Terms: conditions — Polycystic Ovary Syndrome; Menstruation Disturbances; Insulin Resistance; Metabolic Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood serum samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Polycystic ovary syndrome (PCOS)+ insulin resistance (IR)
  Interventions: Diagnostic Test: Measurement of interleukin-6 (il-6) concentration in blood serum; Diagnostic Test: Measurement of fasting tumor necrosis factor α (TNF-α) concentration; Diagnostic Test: Measurement of interleukin-18 (il-18) concentration; Diagnostic Test: Measurement of interleukin-4 (il-4) concentration
- Polycystic ovary syndrome (PCOS)+ no insulin resistance (IR)
  Interventions: Diagnostic Test: Measurement of interleukin-6 (il-6) concentration in blood serum; Diagnostic Test: Measurement of fasting tumor necrosis factor α (TNF-α) concentration; Diagnostic Test: Measurement of interleukin-18 (il-18) concentration; Diagnostic Test: Measurement of interleukin-4 (il-4) concentration
- No PCOS
  Interventions: Diagnostic Test: Measurement of interleukin-6 (il-6) concentration in blood serum; Diagnostic Test: Measurement of fasting tumor necrosis factor α (TNF-α) concentration; Diagnostic Test: Measurement of interleukin-18 (il-18) concentration; Diagnostic Test: Measurement of interleukin-4 (il-4) concentration

INTERVENTIONS:
Diagnostic Test: Measurement of interleukin-6 (il-6) concentration in blood serum — Measurement of fasting interleukin-6 (il-6) concentration in fasting venous blood serum
Diagnostic Test: Measurement of fasting tumor necrosis factor α (TNF-α) concentration — Measurement of fasting tumor necrosis factor α concentration in fasting venous blood serum
Diagnostic Test: Measurement of interleukin-18 (il-18) concentration — Measurement of interleukin-18 (il-18) concentration in fasting venous blood serum
Diagnostic Test: Measurement of interleukin-4 (il-4) concentration — Measurement of interleukin-4 (il-4) concentration in fasting venous blood plasma

SUMMARY:
The study will involve measurements and comparisons of the concentrations of pro-inflammatory cytokines: IL-6, TNF-α, IL-18, as well as anti-inflammatory cytokine IL-4 in women with polycystic ovary syndrome (PCOS) and insulin resistance, women with polycystic ovary syndrome without carbohydrate metabolism disorders, and women without PCOS (control group).

DETAILED DESCRIPTION:
Polycystic ovary syndrome (PCOS) is the most common endocrinopathy among women of reproductive age, which, in addition to menstrual disorders and infertility due to anovulation, is characterized by insulin resistance (IR). The metabolic disturbances associated with PCOS contribute to a higher incidence of cardiovascular diseases and endometrial cancer prior to menopause. The severity of IR in women with PCOS is linked to abdominal obesity. There is an urgent need to identify more precise and universal markers of insulin resistance than the HOMA-IR index or glucose tolerance tests, which are intended to identify existing disorders rather than predispositions. Additionally, there is a need to investigate the balance of pro-inflammatory and anti-inflammatory parameters in PCOS and their relationship with insulin resistance, which is responsible for the development of adverse health complications.

The objective of this study is to measure and compare the concentrations of pro-inflammatory cytokines: IL-6, TNF-α, IL-18, and the anti-inflammatory cytokine IL-4 in women with polycystic ovary syndrome (PCOS) and insulin resistance, women with polycystic ovary syndrome without carbohydrate metabolism disorders, and women without PCOS (control group).

Tests will be conducted using immunoenzymatic methods (ELISA) and the Erba XL biochemical analyzer. The concentrations of the substances under investigation will be measured and compared among the three study groups. Statistical analysis will be performed using SPSS Statistics software.

ELIGIBILITY:
Inclusion Criteria:

* women aged 18-45 years

Exclusion Criteria:

* previous removal of at least one ovary
* treated diabetes of any type
* diagnosed and treated metabolic diseases
* diagnosed and treated autoimmune diseases
* diagnosed and treated autoinflammatory diseases

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: women aged 18-45 years, managed for menstrual irregularities, infertility or for routine check-up
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-01-20 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Il-6 concentration | up to 6 months
  Measurement and comparison of serum interleukin-6 (il-6) concentration expressed in [pg/ml] in three research groups
Il-18 concentration | up to 6 months
  Measurement and comparison of serum interleukin-18 (il-18) concentration expressed in [pg/ml] in three research groups
Il-4 concentration | up to 6 months
  Measurement and comparison of serum interleukin-4 (il-4) concentration expressed in [pg/ml] in three research groups
TNF-α concentration | up to 6 months
  Measurement and comparison of serum tumor necrosis factor α (TNF-α) concentration expressed in [pg/ml] in three research groups

CONTACTS AND LOCATIONS:
Overall Officials: Kazimierz Pityński, Prof., Ph.D., M.D., Study Chair — Jagiellonian University
Locations (1):
- Jagiellonian University, Krakow, Poland